CLINICAL TRIAL: NCT01310712
Title: Use of Oxybutynin for Treating Hyperhidrosis: A Placebo-control Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nelson Wolosker, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Sao Paulo
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-03

CONDITIONS: Hyperhidrosis
Keywords: hyperhidrosis; oxybutynin
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxybutynin (Experimental): patients will receive in the end of the treatment, 10 mg of oxybutynin a day
  Interventions: Drug: Oxybutynin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oxybutynin — 5 mg every 12 hours for 6 weeks
  Arms: oxybutynin
Drug: placebo — placebo twice a day for 42 days.
  Arms: Placebo

SUMMARY:
Video-assisted thoracic sympathectomy (VATS) provides excellent resolution of palmar and axillary hyperhidrosis but is associated with compensatory hyperhidrosis. Low doses of Oxybutynin can be used to treat palmar hyperhidrosis with fewer side effects.

DETAILED DESCRIPTION:
Introduction: Video-assisted thoracic sympathectomy (VATS) provides excellent resolution of palmar and axillary hyperhidrosis but is associated with compensatory hyperhidrosis. Low doses of Oxybutynin can be used to treat palmar hyperhidrosis with fewer side effects.

Purpose: The objective of this study is to evaluate the effectiveness and patient satisfaction with the use of oxybutynin at low doses comparing to placebo for treating palmar hyperhidrosis.

Methods: This is a prospective, randomized and controlled study. From December 2010 to february 2011, 50 consecutive patients with palmar hyperhidrosis were treated with oxybutynin or placebo. Data were collected from 50 patients, and 5 (10,0%) patients were lost to follow-up. During the first week, patients received 2.5 mg of oxybutynin once a day in the evening. From the 8th to the 42nd day, they received 2.5 mg twice a day, and from the 43rd day to the end of the 12th week, they received 5 mg twice a day. All of the patients underwent 2 evaluations: before and after (12 weeks) the oxybutynin treatment, using a clinical questionnaire; and a clinical protocol for quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hyperhidrosis

Exclusion Criteria:

* Glaucoma and pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement of Quality of life in patients with hyperhidrosis with the use of oxybutynin | 6 weeks
  Using a Quality of life protocol we will study if patients with hyperhidrosis using oxybutynin have an improvement in their quality of life

SECONDARY OUTCOMES:
The use of oxybutynin diminishes hyperhidrosis | 6 weeks
  if the use of oxybutynin diminishes hyperhidrosis

CONTACTS AND LOCATIONS:
Overall Officials: WOLOSKER NELSON, Md, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, São Paulo, Brazil